CLINICAL TRIAL: NCT00932763
Title: An Open-Label, Randomized, Two-Way Crossover, Single Dose Study to Evaluate the Bioavailability of the Test Formulation of Amlodipine 10 mg Tablets (Torrent Pharmaceuticals Limited, India) Compared to a 10 mg Dose of Norvasc® (Pfizer, USA) in 22 Fasted, Healthy Adult Subjects
Brief Title: Study to Evaluate the Bioavailability of the Test Formulation of Amlodipine 10 mg Tablets (Torrent Pharmaceuticals Limited) Compared to a 10 mg Dose of Norvasc® (Pfizer) in 22 Fasted, Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Other Study IDs: 20-085-SA
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
MeSH Terms: interventions — Amlodipine

INTERVENTIONS:
Drug: Amlodipine besylate — 10 mg tablets (Torrent Pharmaceuticals, India)
Drug: Norvasc — 10 mg dose (Pfizer, USA)

SUMMARY:
* Objective:

  * The objective of this study was to assess the relative bioavailability of two formulations of immediate release amlodipine 10 mg under fasted conditions, in healthy subjects.
* Study Design:

  * This was an open-label, single-dose, 2-treatment, 2-period, randomized, crossover study.Twenty-two healthy subjects were enrolled. Subjects who successfully completed the screening process checked into the research center the night before first dose. Subjects who continued to meet inclusion/exclusion criteria the morning of dose were assigned a subject number, based on the order in which they successfully completed the screening process and procedures as outlined in the study protocol. Subjects were randomly assigned to a treatment sequence and received two separate single-dose administrations of study medication, one treatment per period,according to the randomization schedule. Dosing days were separated by a washout period of at least 14 days. Subjects received each of the treatments listed below during the two treatment periods following an overnight fast of at least 10 hours: amlodipine by Torrent Pharmaceuticals Ltd. and Norvasc by Pfizer, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male/Female
* Age: 18 - 45 years.
* Volunteer with BMI of 18-27 kg/m2 with minimum of 50 kg weight.
* Volunteers with minimum blood pressure of 110/75 mmHg.
* Healthy and willing to participate in the study.
* Signed Written Informed Consent for Screening and study.
* Medical case history, physical examination, vital signs, laboratory tests and ECG without significant deviations.
* Negative drug of abuse screening test.
* Non-smokers or smoking less than 10 cigarettes a day and willing to refrain from smoking throughout the course of the study.
* No history of medication, prescription or OTC, for at least 2 weeks prior to study drug administration until study Period II completion.

Exclusion Criteria:

* Clinically relevant abnormal physical findings at the screening examination, which would interfere with the objective of the study.
* Clinically relevant abnormalities in the results of the laboratory screening evaluation.
* Clinically relevant ECG abnormalities.
* Habituation of tobacco necessitating uninterrupted tobacco consumption.
* Addiction to alcohol or history of any drug abuse.
* History of kidney or liver dysfunction.
* History of allergy to the test drug or any drug chemically similar to the drug under investigation.
* Administration/Intake of any prescription or OTC medication for two weeks before the study.
* Patients suffering from any chronic illness such as arthritis, asthma etc.
* HIV, HCV, HBsAg positive volunteers.
* Positive test for drugs of abuse screen.
* Subjects suffering from any psychiatric (acute or chronic) illness.
* Administration of any investigational drug in the period 0 to 30 days before entry into the study.
* Intake of barbiturates or any enzyme-inducing drug in last three months.
* History of significant blood loss due to any reason, including blood donation in the past 12 weeks. The total blood loss in last 3 months including anticipated blood loss for this study will exceed 1000 ml.
* History of any bleeding disorder.
* Existence of any surgical or medical condition, which, in the judgement of the clinical investigator, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of volunteers.
* Serious adverse reaction or hypersensitivity to study drug or any of the excipients.
* Inability to communicate or cooperate with the investigator due to language problem, poor mental development or impaired cerebral function.
* Pregnant and nursing mother.
* Female, unless surgically sterile or at least 2 years post-menopausal, not practicing barrier contraceptive methods.
* Contraindications to active or inactive ingredients of the formulation.
* Subject is not willing and able to remain in the study unit for the entire duration of each confinement period and return for all outpatient visits.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- CEDRA Clinical Research, LLC, San Antonio, Texas, United States